CLINICAL TRIAL: NCT06691750
Title: Clinical Impact of Uterine Repair During Cesarean Section with Barbed Suture on the Incidence of Isthmocele and Its Ultrasound and Molecular Characteristics: a Randomized Controlled Trial
Brief Title: Clinical Impact of Uterine Repair During Cesarean Section with Barbed Suture on the Incidence of Isthmocele
Acronym: CESARIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Cristina Mula Navarro, SPECIALIST IN OBSTETRIC AND GYNECOLOGY, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HCB/2024/0196
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Isthmocele; Cesarean Scar Defect; Pelvic Pain; Spotting; Infertility; Uterine Niche; Uterine Abnormal Bleeding; Niche
Keywords: Isthmocele; Uterine niche; Cesarean scar defect; Barbed suture; Cesarean section
MeSH Terms: conditions — Pelvic Pain; Metrorrhagia; Infertility

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, double-blind, two-parallel clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group: Uterine repair with barbed suture (Experimental): Uterine closure following cesarean section is carried out using an unlocked single-layer barbed suture with an endometrium-free technique.
  Interventions: Device: Barbed suture
- Control Group: Uterine repair with conventional smooth suture (Active Comparator): Uterine repair following cesarean section is performed using a conventional smooth polyglactin suture with a continuous single-layer, endometrium-free technique, in accordance with the standard procedure at our center.
  Interventions: Device: Conventional smooth suture

INTERVENTIONS:
Device: Barbed suture — Size 0 barbed absorbable monofilament suture with unidirectional spikes that includes a loop in one of its ends, not requiring knots.
  Arms: Study Group: Uterine repair with barbed suture
Device: Conventional smooth suture — Size 1 smooth multifilament absorbable polyglactin suture.
  Arms: Control Group: Uterine repair with conventional smooth suture

SUMMARY:
Pregnant women, irrespective of their pregnancy risk, who undergo a cesarean section for any reason will be randomized to one of two suturing techniques: conventional suture or barbed suture for uterine repair after the cesarean section. Following surgery, these patients will be followed up for clinical outcomes, ultrasound evaluation of the uterine scar, and study of the hypoxic-inflammatory environment of the uterine cavity.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted among pregnant women, irrespective of their pregnancy risk, undergoing cesarean sections at a tertiary care hospital. Participants will be randomly assigned to one of two groups: the intervention group, which will receive barbed suture for myometrial repair following the cesarean section, or the control group, which will receive conventional smooth suture. This study aims to compare a range of outcomes related to clinical, ultrasonographic, and molecular parameters of the uterine scar and the development of isthmocele.

Main hypothesis: The use of barbed suture for hysterorrhaphy during cesarean section, compared to conventional smooth sutures, results in reduced ischemia and necrosis of the myometrial tissue, facilitating better healing. This is associated with a lower incidence of isthmocele at six months postpartum, and a decrease in its ultrasound dimensions, evaluated by transvaginal ultrasound with hysterosonography.

Secondary hypothesis:

* The use of barbed suture during cesarean delivery leads to a reduction in molecular biomarker levels of hypoxia and inflammation within the uterine cavity.
* The employment of barbed suture is associated with a decrease in the frequency of symptoms related to isthmocele in the short term, or a lower intensity of symptoms if they occur, compared to conventional suture.
* Patients who develop isthmocele after cesarean delivery present predisposing myometrial characteristics and additional risk factors compared to patients with normal healing.
* The study of myometrial texture patterns based on ultrasound images of the uterine wall in the postpartum period following cesarean delivery may provide predictive data regarding the risk of developing isthmocele at six months postpartum.
* The stiffness of the uterine scar measured by the strain ratio (SR) is lower among patients included in the barbed suture group than in patients in the conventional suture group.
* Uterine repair with barbed suture during the cesarean section leads to better perinatal outcomes in the subsequent pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who deliver at Hospital Clinic of Barcelona by a planned, intrapartum or urgent cesarean section, irrespective of their pregnancy risk.
* Had accepted to participate in the study during the third trimester of gestation.
* Patients who accept a 6-month follow-up visit.
* Minimal maternal age of 18 years old.

Exclusion Criteria:

* Patients who end up delivering in another center.
* Patients who deliver by vaginal route.
* Patients diagnosed with isthmocele prior to the current pregnancy.
* Need for histerectomy in the following 6 months after delivery.
* Patients with known allergies to any of the components of the barbed suture.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Isthmocele | Six months after cesarean section.
  Rate of isthmocele six months after cesarean section examined by transvaginal ultrasonography with hysterosonography.
Ultrasonographic Measurements of Isthmocele | Six months after cesarean section.
  Ultrasonographic characteristics of isthmocele measured by niche length, niche depth, niche width, residual myometrial thickness (RMT) and niche size (niche depth/niche depth+RMTx100[%]).

SECONDARY OUTCOMES:
Intrauterine molecular markers of hypoxia and inflammation | Six months after cesarean section.
  Concentrations of the following biomarkers will be assessed by analyzing an endocavitary lavage of the uterus: VEGF-A (an indirect marker of tissue hypoxia associated with angiogenesis and vasculogenesis), G-CSF, IL-1β, IL-6, IL-10, and TNF-α (inflammatory cytokines), as well as HIF1A (hypoxia-inducible transcription factor).
Symptoms | Six months after cesarean section.
  Evaluation of symptoms related to CSD six months after cesarean section, measured as the presence of one or more of the following: prolonged postpartum bleeding, spotting, abnormal menstrual bleeding, dysmenorrhea, pelvic pain and/or dyspareunia.
Risk factors | Through study completion, an average of 2 years.
  Collection of individual data in relation to the patient characteristics and the surgical procedure to evaluate potential risk factors.
  Individual data: Age at inclusion, ethnicity, educational level, parity, number of cesarean deliveries, history of uterine surgery or other abdominal surgeries, body mass index, smoking status, gestational or pregestational diabetes, hypertension, other medical conditions.
  Surgical data: Location of the hysterotomy, need for additional hemostatic sutures, need for hemostatic material at the surgical site, requirement for antifibrinolytic or uterotonic treatment to control bleeding, estimated blood loss during the surgery.
Ultrasonographic myometrial texture patterns | Six months after cesarean section.
Stiffness of the uterine scar | Six months after cesarean section.
  Stiffness differences of the uterine scar between the two groups will be compared by measuring the strain ratio (SR).
Perinatal outcomes in following pregnancies | Through study completion, an average of 4 years.
  Perinatal outcomes in subsequent pregnancies will be measured as the presence of one of the following: miscarriage, ectopic pregnancy, uterine rupture, placental accretism, cesarean delivery among others.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No